CLINICAL TRIAL: NCT01133028
Title: Classroom-Level Intervention to Promote Peers' Acceptance of Children With Attention-Deficit/Hyperactivity Disorder (ADHD)
Brief Title: Classroom-Level Intervention to Promote Peers' Acceptance of Children With Attention Deficit Hyperactivity Disorder (ADHD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Amori Y Mikami, Assistant Professor, University of Virginia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0066-00
Record Dates: First submitted 2010-05-10; First posted 2010-05-28 (Estimated); Last update posted 2010-05-28 (Estimated); Status verified 2010-05

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention Deficit Hyperactivity Disorder (ADHD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combined (Experimental): This represents a combination of the tolerance training and behavioral management interventions together.
  Interventions: Behavioral: Behavioral contingency management; Behavioral: Tolerance training
- Behavioral management (Active Comparator): This represents the behavioral contingency management intervention only.
  Interventions: Behavioral: Behavioral contingency management

INTERVENTIONS:
Behavioral: Behavioral contingency management — Teachers will learn to use reinforcements and response cost procedures to encourage children's display of prosocial behaviors.
Behavioral: Tolerance training — Teachers will be instructed in procedures to encourage the peer group to be accepting of children with ADHD.
  Arms: Combined

SUMMARY:
Children with Attention-Deficit/Hyperactivity Disorder (ADHD) comprise about 5-10% of the elementary school-age population. One place where children with ADHD have great difficulty is in being accepted by peers and in making friends. It has unfortunately been very difficult for the field to find good treatments for peer relationship problems for this population. Even when children with ADHD do improve their behavior, it is common that peers do not seem to like the child with ADHD any better. This may happen because children often have negative reputations with their classmates that are hard to change. That is, once a class of children get the impression that one child is disliked or the social outcast, even if that child's ADHD symptoms get better, the peer group may not notice any of these improvements. It is hypothesized that the elementary school teacher may be able to help peers notice positive behavior changes in children with ADHD when they do occur. This clinical trial will design and pilot-test an intervention that would train teachers in classroom practices to reduce the peer rejection of students with ADHD. The pilot test will be conducted in a summer program created to be similar to a regular school classroom in structure. If the treatment seems to succeed in the summer program, then it will be tried in regular classrooms in a future study.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 6-8
* Primary diagnosis of ADHD

Exclusion Criteria:

* Pervasive Developmental Disorder
* Verbal IQ below 75

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 102 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-09 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Child Peer Relationships | The first day of the treatment and the last day of the treatment (two weeks later)
  This is collected in the summer program in which the intervention will be adminstered. On the first day of the program (before treatment begins), pre-test measures will be taken. They will be re-taken on the last day of the program two weeks later (on the last day of treatment). Peer relationships will be assessed by peer sociometric interviews. Proportion scores of peer acceptance, reciprocated friendship, and inclusion in social networks will be calculated, and changes in these outcomes over the summer prorgam will be considered as evidence to evaluate the treatment.

SECONDARY OUTCOMES:
Child Behavior Problems | The first day of the treatment and the last day of the treatment (two weeks later)
  This measure will be collected on the same time frame as is the primary outcome measure. Children's behavior problems (aggression, inattention, hyperactivity/impulsivity, social withdrawal) will be assessed by teacher report and by observation. Changes in behavior problems during this period will be considered as evidence for the efficacy of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Amori Y Mikami, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States